CLINICAL TRIAL: NCT06536894
Title: The Effect of the Presence Fibromyalgia Syndrome on Anthropometric and Ultrasonographic Measurements in Obstructive Sleep Apnea Syndrome
Brief Title: Fibromyalgia Syndrome on Anthropometric and Ultrasonographic Measurements in Obstructive Sleep Apnea Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Assosc Prof, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEK_2024-12/95
Record Dates: First submitted 2024-07-11; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia Syndrome; Obstructive Sleep Apnea Syndrome
Keywords: Sleep Disorder; Obstructive Sleep Apnea Syndrome; Fibromyalgia Syndrome; anthropometric measurement; ultrasonographic measurement; Polysomnography
MeSH Terms: conditions — Fibromyalgia; Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fibromyalgia syndrome and obstructive sleep apnea: Fibromyalgia patients who were diagnosed with OSAS as a result of polysomnographic examination
- Fibromyalgia syndrome: Fibromyalgia patients who were not diagnosed with OSAS as a result of polysomnographic examination
- Obstructive sleep apnea syndrome.: Patients diagnosed with OSAS as a result of polysomnographic examination and without fibromyalgia

SUMMARY:
Obstructive type sleep apnea syndrome is a clinical condition characterized by apnea, hypopnea and oxygen desaturation due to narrowing of the upper airway during sleep. Obesity is considered a major predisposing factor for OSAS. In addition, various recent studies have reported that various anthropometric measurements such as neck circumference, waist circumference, hip circumference, waist-hip ratio, neck-waist circumference ratio change (increase) in OSAS patients.

DETAILED DESCRIPTION:
Fibromyalgia is a common health problem that is characterized by pain in various parts of the body and is very difficult to diagnose and treat. It affects 2-4% of the population and is more common in women. The presence of OSAS in fibromyalgia patients is more common than in the normal population. There are also common additional symptoms such as excessive daytime sleepiness and delayed sleep latency.

Although it has been reported that the presence of OSAS is more common in fibromyalgia patients, there is no study on the presence of anthropometric measurements, especially neck circumference, that are accepted in OSAS.

The aim of this study is to compare the anthropometric and ultrasonographic measurements of female OSAS patients with and without fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years old
* Being diagnosed with fibromyalgia and having applied to the sleep disorders outpatient clinic or being followed up with the diagnosis of OSAS in the sleep disorders outpatient clinic.
* Agree to participate in the study

Exclusion Criteria:

* Patients under 18 years of age
* Male patients
* Not agreeing to participate in the study
* Neurological diseases that may cause OSAS such as stroke, Parkinson's disease, multiple sclerosis
* Rheumatological, oncological and hematological diseases
* Central type obstructive sleep apnea syndrome
* Thyroid pathology that affects neck circumference measurement

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In order to eliminate gender-based factors
Study Population: Female patients diagnosed with fibromyalgia who applied to the sleep disorders outpatient clinic operating within the Department of Neurology and underwent polysomnography with sleep problems, as well as patients diagnosed with OSAS, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Measurements | Day 0 ( Baseline)
  Anthropometric measurements will be taken for all patients. These measurements include neck circumference, waist circumference, hip circumference, and with these data, waist-hip ratio and neck-waist circumference ratio will be calculated. Measurements will be made with a tape measure and with patient consent.
Polisomnografi- SLEEP LATENCE | Day 0 ( Baseline)
  Sleep latency time will be measured in polysomnography
Polisomnografi -SLEEP ACTIVITY | Day 0 ( Baseline)
  Sleep efficiency will be measured during polysomnography
Polisomnografi -REM time | Day 0 ( Baseline)
  REM time will be measured in minutes during polysomnography
Polisomnografi -NREM STAGES | Day 0 ( Baseline)
  During polysomnography, NREM stages will be measured at 1 min, 2 min, and 3 min.
Polisomnografi - NUMBERS OF APNE | Day 0 ( Baseline)
  Numbers of apnea will be recorded in polysomnographic measurements.
Polisomnografi -NUMBER OF HYPOPNEA | Day 0 ( Baseline)
  Numbers of hypopnea will be recorded in polysomnographic measurements
Polisomnografi -Apnea hypopnea index (AHI) in polysomnography; Apnea hypopnea index (AHI) will be evaluated on a supine, non-supine basis. | Day 0 ( Baseline)
  Apnea hypopnea index (AHI) will be evaluated in polysomnography.According to the AHI level; It will be classified as SIMPLE SNORING (AHİ<5), LIGHT OSAS (AHİ 5-15), MEDIUM OSAS (AHİ 15-30), HEAVY OSAS (AHİ 30+ )
Polisomnografi-REM | Day 0 ( Baseline)
  REM times will be evaluated in polysomnography
Polisomnografi-NonREM | Day 0 ( Baseline)
  NonREM times will be evaluated in polysomnography
Polisomnografi -Apnea hypopnea index (AHI) REM, NONREM in polysomnography; Apnea hypopnea index (AHI) will be evaluated on a supine, non-supine basis. | Day 0 ( Baseline)
  Apnea hypopnea index (AHI) will be evaluated as REM, NONREM, Supine, non-supine in polysomnography.According to the AHI level; It will be classified as SIMPLE SNORING (AHİ<5), LIGHT OSAS (AHİ 5-15), MEDIUM OSAS (AHİ 15-30), HEAVY OSAS (AHİ 30+ )
Polisomnografi -OXYGEN DESATURATION INDEX | Day 0 ( Baseline)
  Minimum oxygen saturation and average oxygen saturation will be measured in polysomnography.
submental ultrasonography | Day 0 ( Baseline)
  All patients will undergo submental ultrasonography to measure tongue base thickness and lateral pharyngeal wall thickness.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Day 0 ( Baseline)
  The Pittsburgh Sleep Quality Index will be used to evaluate sleep quality. The survey consists of 21 questions and a high score indicates poor sleep quality.
Fibromyalgia Impact Scale | Day 0 ( Baseline)
  The fibromyalgia levels of the participants will be evaluated with the Fibromyalgia Impact Scale. High scores indicate increased disease activity. Consists of 10 questions Maximum score is 80. Turkish validity and reliability was done

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Assoc. Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mutlu P, Zateri C, Zohra A, Ozerdogan O, Mirici AN. Prevalence of obstructive sleep apnea in female patients with fibromyalgia. Saudi Med J. 2020 Jul;41(7):740-745. doi: 10.15537/smj.2020.7.25165. PMID 32601643
- [Background] Cigdem Karacay B, Sahbaz T, Zerman N, Tuncay F. The impact of fibromyalgia syndrome on obstructive sleep apnea syndrome in terms of pain threshold, daytime symptoms, anxiety, depression, disease severity, and sleep quality: a polysomnographic study. Sleep Breath. 2023 Aug;27(4):1473-1479. doi: 10.1007/s11325-023-02831-2. Epub 2023 Apr 18. PMID 37071285
- [Background] Mohan Lal B, Vyas S, Malhotra A, Ray A, Gupta G, Pandey S, Pandey RM, Aggarwal S, Sinha S. Ultrasonography of the neck in patients with obstructive sleep apnea. Sleep Breath. 2023 Jun;27(3):903-912. doi: 10.1007/s11325-022-02682-3. Epub 2022 Jul 23. PMID 35871215
- [Background] Deng H, Duan X, Huang J, Zheng M, Lao M, Weng F, Su QY, Zheng ZF, Mei Y, Huang L, Yang WH, Xing X, Ma X, Zhao W, Liu X. Association of adiposity with risk of obstructive sleep apnea: a population-based study. BMC Public Health. 2023 Sep 21;23(1):1835. doi: 10.1186/s12889-023-16695-4. PMID 37735660